CLINICAL TRIAL: NCT02576340
Title: Spasmolytic (Otilonium Bromide) Use in Upper Gastrointestinal Endoscopy: Randomized Prospective Trial
Brief Title: Spasmolytic in Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, barış sevinç, M. D., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ob002
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Gastroscopy
MeSH Terms: interventions — octylonium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (Active Comparator): drug was administered
  Interventions: Drug: otilonium bromide
- control (No Intervention): no drug administered

INTERVENTIONS:
Drug: otilonium bromide — otilonium bromide was administered before the procedure
  Arms: study

SUMMARY:
Upper gastrointestinal system endoscopy is widely used for diagnostic approach. To increase the tolerability and compliance of the patient, sedation is applied. There are many studies showing that sedation increases the patient compliance and the tolerability. However, spasmolytic use in GE has not been evaluated yet.

ELIGIBILITY:
Inclusion Criteria:

* no hypersensitivity to the agent.

Exclusion Criteria:

* Emergent cases,the cases with low mental compatibility and pregnant women were excluded from the study. Moreover, the procedures under sedation, cases with disorders decreasing the intestinal motility like hypothyroidism and diabetes were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
motility | 3 months
  decrease in motility during the procedure (number of peristaltic moves in a minute)

SECONDARY OUTCOMES:
patient tolerance | 3 months
  patient tolerance will be determined by questionnaire